CLINICAL TRIAL: NCT03014531
Title: Daily Almond Intake as a Preload Before Meals Versus as a Snack Between Meals Has Different Effects on Body Fat Percentages and the Lipid Profile in a Randomized Controlled Trial of Young Adults in South Korea
Brief Title: Effects of Daily Almond Intake as a Preload Before Meals Versus as a Snack Among Korean Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ICAN Nutrition Education and Research (Industry)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-KIMH-01-ICAN
Record Dates: First submitted 2016-12-25; First posted 2017-01-09 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Adult Young and Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- almond (Experimental): In this group, participants were provided with 56 g of almonds per day either as preload before meals or snack between meals. A snack was defined as an eating event that occurred between participants' regular meals, specifically two hours before and after meals. All the participants in almond group were provided daily portions of packaged almonds.
  Interventions: Other: almond
- high-carbohydrate control food item (Other): In this group, participants were provided with high-carbohydrate control food item that had a similar number of calories as 56 g of almonds.
  Interventions: Other: high-carbohydrate control food

INTERVENTIONS:
Other: almond
  Arms: almond
Other: high-carbohydrate control food
  Arms: high-carbohydrate control food item

SUMMARY:
The study was conducted to investigate the effects of daily almond intake based on the timing of almond consumption (i.e., almond consumption as a preload or between-meal snack) on body composition, lipid profile, and oxidative and inflammation indicators among young Korean adults.

DETAILED DESCRIPTION:
The current study was conducted to investigate the effects of daily almond intake on body composition, lipid profile, and oxidative and inflammation indicators among young Korean adults based on the timing of almond consumption. Participants were randomly assigned to one of three groups: (1) a pre-meal group (PM; n = 58) in which participants were instructed to consume 56 g of almonds per day as a preload when having regular meals; (2) a snack group (SN; n =55) in which participants were instructed to consume 56 g of almonds between meals as snacks; and (3) a control group (CL; n = 56) in which participants were provided high-carbohydrate iso-caloric control food. The three-day diet records, including two consecutive weekdays and one weekend day, were done once before the trial and twice during the trial. Body composition was assessed through multi-frequency whole-body bioimpedance measurement using InBody 620 (Biospace Co., Ltd, Seoul, Korea).After a 12-hour fast, blood samples were taken at the baseline time point (week 0) and at weeks 8 and 16 by standard venipuncture. The serum total cholesterol and triglycerides levels were measured by the enzymatic-colorimetric method using a Cobas 8000 c702 chemistry analyzer (Roche Diagnostics; Mannheim, Germany). HDL cholesterol and LDL cholesterol levels were determined via homogeneous enzymatic colorimetry.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers
* age 20-39 yr
* Male and Female non-smokers
* BMI 17-30 kg/m2
* under Korean habitual diet

Exclusion criteria:

* any diseases
* any weight change 6 mo before the study
* >2 times/wk nut consumption
* frequent alcohol consumption
* any use of nutrient supplements
* erratic exercise habits
* women who were with irregular menses, taking birth control pills, pregnant or lactating

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes of body fat percentages from baseline | week 8
Changes of blood lipid profiles from baseline | week 8
Changes of body fat percentages from baseline | week 16
Changes of blood lipid profiles from baseline | week 16
Changes of body fat percentages from baseline | week 20
Changes of blood lipid profiles from baseline | week 20

SECONDARY OUTCOMES:
Changes of blood IL-6 levels | week 8
Changes of blood IL-6 levels | week 16

CONTACTS AND LOCATIONS:
Locations (1):
- ICAN Nutrition Education and Research, Seoul, South Korea

REFERENCES:
- [Derived] Liu Y, Hwang HJ, Ryu H, Lee YS, Kim HS, Park H. The effects of daily intake timing of almond on the body composition and blood lipid profile of healthy adults. Nutr Res Pract. 2017 Dec;11(6):479-486. doi: 10.4162/nrp.2017.11.6.479. Epub 2017 Nov 22. PMID 29209458